CLINICAL TRIAL: NCT00590083
Title: Administration of Virus-Specific Cytotoxic T-Lymphocytes for the Prophylaxis and Therapy of Adenovirus Infection Post Allogeneic Stem Cell Transplant
Brief Title: Administration of Virus-Specific Cytotoxic T-Lymphocytes
Acronym: LYPTAIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, catherine bollard, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14097-LYPTAIST; NCT00111033 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-10 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Adenovirus Infection
Keywords: stem cell transplantation; adenovirus; Cytotoxic T-Lymphocytes; prophylaxis
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Virus Specific Cytoxic T lymphocytes (Experimental): Virus Specific Cytoxic T lymphocytes
  Interventions: Biological: CTL administration

INTERVENTIONS:
Biological: CTL administration — Adenovirus specific T cells will be given by intravenous injection from day 30 post transplant.
  One infusion of Adenovirus-specific CTL given to patients at risk for Adenoviral disease after matched or mismatched unrelated or matched or mismatched related donor stem cell transplant. Four dose levels will be explored. The lowest level will be 1x dose of 5x10e6cells/m2 and the highest will be 1x dose of 1.35x10e8/m2.

SUMMARY:
The main purpose of this study is to see if these T-lymphocytes are safe. To make these Ad-specific T lymphocytes the investigators will obtain blood from the stem cell donor and transfer Ad into another type of blood cell, called monocytes. These cells can then stimulate the T lymphocytes and train them to kill cells infected with Ad. The investigators will then grow these Ad-specific T lymphocytes by more stimulation with Ad-infected monocytes and a third type of blood cell called a B lymphoblast from the donor. After testing the T -lymphocytes, the investigators will inject them into patients after transplant who are at high risk of serious Ad virus infection. The investigators will make sure the injected cells are safe and see if they affect the growth and behavior of adenoviruses in the patient's own body.

DETAILED DESCRIPTION:
Viral infection is one of the major causes of morbidity and mortality in patients who receive bone marrow transplantation (BMT) from unrelated or mismatched donors. This increased risk of infection relates to a number of factors including the immunosuppressive regimens these patients receive, delayed immune recovery and the greater genetic disparity between donor and recipient that result in defective interactions between antigen presenting cells and immune system effector cells. In most cases viral infection post BMT results from reactivation of latent virus and CMV, EBV and adenoviruses (Ad) are the commonest viral pathogens causing disease after transplant.

The incidence of Ad infection is >25% for patients at risk in the first 100 days after transplant 1 2. In the transplant population, adenovirus is recoverable from many sites and may cause hemorrhagic cystitis, pneumonitis, nephritis, hepatitis, colitis and pancreatitis, often with severe morbidity and a mortality approaching 60%3. The most frequently used drug for the treatment of adenoviral infections is Cidofovir. But while there are occasional reports of responses to Cidofovir, no approved antiviral agent has proven efficacy for the treatment of severe Ad disease, nor are there any prospective randomized, controlled trials of potentially useful anti-Ad therapies 4. With the increasing use of so-called submyeloablative or reduced intensity, highly immunosuppressive conditioning regimens, higher rates of Ad infections/reactivation have been observed due to prolonged immune suppression. The onset of Ad disease/reactivation has recently been reported to occur at a median of 18 days post-transplant (range -7/>+100) 2.

As viral complications in these patients are clearly associated with the lack of recovery of virus-specific cellular immune responses, reconstitution of the host with in vitro expanded CTLs is an effective approach to prevent and treat these diseases. Adoptive immunotherapy with in vitro expanded CTLs has proved effective in preventing and treating diseases related to Epstein Barr virus (EBV) infections 5; 6 and cytomegalovirus (CMV) reactivations7 in hematopoietic stem cell transplant (HSCT) recipients. A promising strategy to generate donor-derived Ad-specific CTL is the infection of monocytes that direct the CTL response to viral capsid antigens8. This approach allows exposure to all proteins in the Ad protein coat, leading to presentation of multiple, undefined antigen epitopes. Hence, the investigators now plan to use a recombinant Ad vector for infection of donor-derived monocytes. These infected monocytes will then be used as antigen presenting cells (APC) to generate Ad-specific CTL in vitro. For the expansion of the Ad-specific CTL, the second stimulation will use irradiated, Ad-infected monocytes and subsequent stimulations will use donor-derived Lymphoblastoid Cell Lines (LCL) transduced with the Ad vector as an APC 9.

The investigators propose to evaluate this approach for the prophylaxis of Ad reactivation and disease in the recipients of matched unrelated donor or mismatched family member bone marrow allografts, who are at high risk for this complication. Initially, the investigators will give the donor-derived Ad-specific CTLs to patients in a dose escalation study to determine their safety and immunologic and virologic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic (i.e. HLA matched or mismatched related or unrelated) donor stem cell transplants at risk for Adenoviral disease
* No evidence of GVHD > Grade II at time of enrollment
* Life expectancy > 30 days
* No severe intercurrent infections
* Lansky/Karnofsky scores >60
* Absence of severe renal disease (Creatinine > x 3 normal for age)
* Absence of severe hepatic disease (direct bilirubin > 3 mg/dl or SGOT > 500)
* Patient must be at least 30 days post transplant to be eligible to receive CTL
* Not receiving Cidofovir
* Patient has not received other viral specific CTL prophylactically within 4 weeks of receiving Adv-CTL
* Patient/guardian able to give informed consent

Exclusion Criteria:

* Patients with GVHD Grades III-IV
* Patients with hepatic or renal disease as specific above
* Patient has received other viral specific CTL (e.g. EBV-specific CTL or CMV-specific CTL) within 4 weeks of receiving Adv-CTL
* Patients with Adenoviral disease prior to day +30 post transplant Adenoviral diseases defined as the presence of more than two sites positive for adenovirus by culture
* Patients with less than 50% donor chimerism in either peripheral blood or bone marrow or patients with relapse of original disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
safety, toxicity and MTD of 1 IV injection of donor-derived adenovirus-specific CTLs given as adenovirus prophylaxis to patients at risk of developing adenovirus infection after allogeneic stem cell transplant. | 1 year
To evaluate the recovery of virus-specific immunity after CTL infusion and assess its correlation with protection from viral load and disease. | 1 year
To obtain preliminary information regarding whether the presence of antigen is required for Ad-specific CTL persistence in vivo. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bollard, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - National Institute of Health (NIH), Washington D.C., District of Columbia
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Leen AM, Christin A, Myers GD, Liu H, Cruz CR, Hanley PJ, Kennedy-Nasser AA, Leung KS, Gee AP, Krance RA, Brenner MK, Heslop HE, Rooney CM, Bollard CM. Cytotoxic T lymphocyte therapy with donor T cells prevents and treats adenovirus and Epstein-Barr virus infections after haploidentical and matched unrelated stem cell transplantation. Blood. 2009 Nov 5;114(19):4283-92. doi: 10.1182/blood-2009-07-232454. Epub 2009 Aug 21. PMID 19700662